CLINICAL TRIAL: NCT06011655
Title: Attitudes and Stigma Towards Suicidal Behavior in Intensive Care and Emergency Service Nurses
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: SBU-NK-02
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-08

CONDITIONS: Suicide; Stigma, Social
Keywords: suicide; stigma
MeSH Terms: conditions — Suicide; Social Stigma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General intensive care and emergency servise nurses: The research was planned as a descriptive study to be carried out in the general intensive care and emergency departments of the Sanatorium Hospital. After obtaining permission from the institution where the study will be conducted, the "Personal Information Form", "Attitude Towards Suicide Attempts" and "Stigma towards Suicide" scale will be sent to the nurses working in the general intensive care and emergency services of the hospital by the researcher online via Google Forms. Nurses, 5-10 min to answer. They will fill in the scales, which will continue, on their duty leave or on holidays.

SUMMARY:
The aim of this study is to determine the attitudes and stigmatization levels of nurses working in the intensive care and emergency departments towards suicidal behavior.

DETAILED DESCRIPTION:
Suicide is an important and priority public health problem. In the last 45 years, the suicide rate in the world has increased by 60%. About 800,000 people die each year due to suicide. Suicide can be prevented with timely, evidence-based, and often low-cost interventions. The first places that individuals who attempt suicide apply are often the emergency departments of hospitals. These individuals are then referred to intensive care units for close follow-up of physical findings and treatment according to the results of the suicide attempt. Nurses working in the emergency room and general intensive care unit should consider the need for psychosocial support while taking precautions against the physiological consequences of suicide in order for the individual to survive. In the care of an individual who has attempted suicide, the nurse has responsibilities such as providing education to the patient, creating a safety plan, counseling for the restriction of deadly vehicles, quick referral to the necessary places, and providing contact with post-discharge care. It is a priority in the care of the individual that the nurse reduces the sense of hopelessness of the individual who comes with a suicide attempt, re-establishes the sense of commitment to other people, increases compliance with the treatment, motivates for change, and establishes therapeutic communication. In this regard, the knowledge level of healthcare professionals and nurses who provide primary care to patients, and their attitudes towards suicide are important. When the literature is examined, studies on the attitudes of health professionals working in the emergency room toward suicide attempts have been observed, but no research has been found that determines both the attitudes and stigmatization levels of intensive care and emergency room nurses toward suicidal behavior. For this reason, this study was planned to determine the attitudes and stigmatization levels of nurses working in the general intensive care and emergency departments towards suicidal behavior.

ELIGIBILITY:
Inclusion Criteria:

* Having no barriers in oral and written communication in Turkish
* Volunteering to participate in research
* Working in the general intensive care or emergency department of the hospital

Exclusion Criteria:

* Giving incomplete or incorrect information to forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer nurses working in the general intensive care and emergency departments of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Attitude towards suicidal behavior | 5 months, the scale will be filled in once.
  It will determine the level of stigmatization of the nurses towards the suicidal behavior of individuals. In the measurement "Suicidal Stamping Scale" will be used. The highest score that can be obtained from the scale is 140 and the lowest score is 28. from scale A high score indicates a positive attitude.

SECONDARY OUTCOMES:
Stigmatization of suicidal behavior | 5 months, the scales will be filled in once.
  It will determine the attitudes of nurses towards the suicidal behavior of individuals. "Attitude Scale Towards Attempted Suicide" will be used in its measurement. The scale does not have a total score. Stigma bottom of the scale High scores from the sub-dimension indicate high stigma towards suicide, high scores from the isolation/depression sub-dimension indicate that suicide is more associated with depression and isolation.
  High scores from the glorification/normalization subscale indicate that suicide is considered normal or that people who commit suicide are glorified.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Yüksel, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Sağlık Bilimleri University, Ankara, Turkey (Türkiye)